CLINICAL TRIAL: NCT05457179
Title: Physical Activity to Reduce Cardiometabolic Risk in Adults With Serious Mental Illness (PARCS) Study
Acronym: PARCS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: Augusta University (Other); Dartmouth College (Other); University of Cincinnati (Other)
Responsible Party: Principal Investigator, Gina Besenyi, Assistant Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11008
Record Dates: First submitted 2022-03-19; First posted 2022-07-13 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Mental Disorders, Severe; Mental Illness Persistent
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm multi-site randomized clinical trial. The intervention arm will consist of peer counselor-led park-based physical activity sessions 3 days per week for 12 weeks incorporated into weekly peer counseling sessions. The active control arm will consist of physical activity and park information. Both arms will include standard of care peer-group counseling services.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): PARCS is a park-based physical activity intervention including aerobic and resistance training adapted for adults with serious mental illness and led by certified peer counselors as part of peer group mental health recovery services.
  Interventions: Behavioral: Park-based physical activity
- Active Control (Active Comparator): The active control group will receive information about the importance of park-based PA and a map of local park locations but will not participate in structured park-based PA sessions. Participants in the control group will be invited to participate in park PA sessions after they have completed posttest.
  Participants in both groups will receive usual care outpatient peer group treatment services, including routine counseling and health and wellness information/activities given by CPSs.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Park-based physical activity — The experimental arm will optimize a 12-week intervention 3 days/wk, last approximately 60 minutes, and consist of 10 minutes of warm up, 15 minutes of simple strength training activities, 25 minutes of moderate to vigorous aerobic activities (e.g., walking), and 10 minutes of cool down. The eight full-body strength training exercises will use body weight and/or elastic bands and will include a circuit of chest press, seated row, squat, shoulder press, biceps curl, triceps extension, calf raise, and reverse crunch. Sessions will include education and skill building activities focused on Social Cognitive Theory mechanisms of change including self-efficacy, goal setting, and social support. Under the guidance of trained research staff, certified peer specialists who have experience working with peer groups, will be selected to help deliver the intervention.
  Arms: Intervention
Behavioral: Active Control — The active control group will receive information about the importance of park-based PA and a map of local park locations but will not participate in structured park-based PA sessions. Participants in the control group will be invited to participate in park PA sessions after they have completed posttest.
  Arms: Active Control

SUMMARY:
The aim of this project is to trial the protocol of a park-based physical activity (PA) intervention in adults with serious mental illness (SMI) in a community mental health center's peer support program.

DETAILED DESCRIPTION:
Adults with serious mental illness or serious mental illness (SMI) suffer from drastically higher rates of premature mortality (as much as a 10-25 years reduction in life expectancy) compared to the general population. Co-morbid medical conditions (i.e., heart disease, diabetes) are a fundamental cause. The iatrogenic cardiometabolic effects associated with antipsychotic drugs complicate matters. Underlying modifiable cardiometabolic risk factors (e.g., obesity, hypertension, poor physical fitness) are more prevalent and manifest earlier in the lifecourse in persons with SMI compared with the rest of society. Physical activity (PA) is an extensively recognized modifiable behavior that can reduce numerous cardiometabolic risk factors as well as improve quality of life (QOL) in people with SMI. Evidence-based methods for developing PA interventions among adults with SMI often incorporate individual attention, peer counselors, structured group PA, novel technology, self-monitoring, and behavior change strategies. However, challenges exist for both delivery and sustainability of effective PA treatment strategies for people with SMI in community settings. Indeed, development and testing of innovative, evidence-based PA interventions with SMI populations has been identified as a top research priority.

Parks are acknowledged as key community PA intervention settings given their low cost, ubiquity, and provision of structured and unstructured PA opportunities. Parks offer numerous physical, psychological, and social benefits associated with improved health behaviors and outcomes. Growing evidence, including our own, has documented relationships between access and use of parks and green space with greater PA, mood, and QOL, and less obesity, stress, morbidity and mortality. Further, outdoor PA is associated with increased enjoyment, satisfaction, and long-term adherence to PA, supporting it as an ideal approach to PA behavior change, especially among those with SMI. Despite potential benefits of park-based PA, few interventions have been tested rigorously, and none have focused specifically on adults with SMI. Certified peer specialists (CPSs), trained persons with lived recovery experience working in mental health settings, offer a potential delivery mechanism for park-based PA. Pulling from the Recovery Model incorporating elements of peer support and collaborative treatment approaches our long-term goal is to maximize the reach and clinical impact of evidence-based PA interventions to reduce cardiometabolic risk among adults with SMI through the use of existing CPS services and park-based PA.

The PARCS Study uses a novel approach for physical activity (PA) intervention delivery and sustainability among adults (18+yrs) with SMI through incorporation of freely available park resources into established peer counseling programs. The purpose of the PARCS study is two-fold: 1) Test the feasibility and acceptability of a CPS-led PA intervention among adults with SMI in park settings, and 2) evaluate the effectiveness of the PARCS intervention on a) SCT mechanisms of action (i.e., PA self-efficacy, goal setting, and social support) and b) PA, fitness, and health outcomes.

The PARCS Study aims to establish a sustainable, scalable, and reimbursable intervention model by leveraging existing resources (CPS services, parks) to reduce cardiometabolic risk in adults with SMI. Combining information from previous feasibility and effectiveness PA trials with adults with SMI, park-based PA literature, qualitative and quantitative feedback from pilot studies, the PARCS Study will optimize a 12-week PA intervention originally developed for people with chronic schizophrenia in an indoor setting, to an outdoor group exercise setting in parks. This study will utilize a two-arm randomized active control group design with pre- and posttest measures (n=100). Arm one, will consist of a 12-week park-based PA intervention, including sessions three days per week at times and days convenient for each participating facility. Under the guidance of trained research staff, four CPSs, who have experience working with peer groups, will be selected to help deliver the intervention. Park-based activity sessions will last approximately 60 minutes and consist of 10 minutes of warm up, 15 minutes of simple strength training activities, 25 minutes of moderate to vigorous aerobic activities (e.g., walking), and 10 minutes of cool down. The eight full-body strength training exercises will use body weight and/or elastic bands and will include a circuit of chest press, seated row, squat, shoulder press, biceps curl, triceps extension, calf raise, and reverse crunch. These activities have been selected to improve functional capacity of common daily living activities (e.g., ability to stand from seated position, lift groceries, use stairs, etc). During pilot studies, an ACSM-certified group fitness instructor developed scaled group-based activity sessions that progress in activity level over time with participants' capabilities. Sessions will strive to incorporate fun, social, adaptable activities that enable a wide variety of subjects to participate. Arm two, the active control group, will receive information about the importance of park-based PA, and a map of park locations but will not participate in park-based PA sessions. Participants in the control group will be invited to participate in park PA sessions after they have completed posttest. Participants in both groups will receive a Fitbit and usual care outpatient peer group treatment services, including routine counseling and health and wellness information/activities given by CPSs.

ELIGIBILITY:
Inclusion Criteria:

* Authorized for peer group treatment through the behavioral health facility
* Medically cleared to participate in physical activity (if indicated by ACSM 11th Edition pre-exercise participation screener)

Exclusion Criteria:

* Under 18 years of age
* Unable to obtain physician clearance (if indicated by ACSM 11th Edition pre-exercise participation screener)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Attendance | Ongoing during the 12-week intervention period
  Feasibility will be assessed by attendance at park PA sessions. Higher attendance indicates greater engagement with the intervention
Acceptability - Change in PA Enjoyment | post 12-week intervention
  Acceptability will be assessed via PA enjoyment captured using the Physical Activity Enjoyment Scale (PACES), an 18-item scale where participants rate feelings about PA on a 7-point Likert scale, from 1 (I enjoy it) to 7 (I hate it).
Acceptability - PA session satisfaction | post 12-week intervention
  Acceptability will also be assessed via PA session satisfaction measured using the abbreviated Physical Activity Class Satisfaction Questionnaire (PACSQ) which rates satisfaction of park-based class sessions on an 8-point Likert scale. PACSQ is a valid measure for capturing client satisfaction within exercise classes in the following nine dimensions: mastery experiences, cognitive development, teaching, normative success, interaction with others, fun and enjoyment, improvement of health and fitness, diversionary experiences, and relaxation. Each of the dimensions of satisfaction is measured using an 8-point Likert scale, with responses ranging from 1="No satisfaction" to 8="Very satisfying". PACSQ has shown acceptable reliability in each of its subscales (all α's ≥ .85), and survey items are highly correlated with participants' intentions to attend a similar course in the future.

SECONDARY OUTCOMES:
Change in Self-efficacy for Exercise | pre and post 12-week intervention
  The SCT mechanism of self-efficacy will be measured using the Self Efficacy for Exercise (SEE) Scale, a 9-item self-report Likert scale asking how confident participants are they could exercise three times a week for 20 minutes under various conditions (felt stressed, felt tired). Answers range from 1 (not confident) to 10 (very confident). The SEE scale has an internal consistency of 0.92 and has been used in a variety of populations.
Change in Self-efficacy and Intensions for Spending Time in Nature | pre and post 12-week intervention
  Self-efficacy and intentions for spending time in nature will be assessed using the Spending Time in Nature Measures, which has high internal consistency (α = .93 self-efficacy; .91 intentions). Self-efficacy will be assessed with 14 items asking participants how confident they are spending at least 2 hours/week in green and natural spaces on a scale from 1 (not confident at all) to 5 (extremely confident). Intensions to spend time in nature will be measured with 8 items asking participants their intentions to spend time in nature in the next three months. Answers are assessed on a 5pt Likert scale where 1 = 'Strongly disagree' to 5 = ' Strongly agree'. The scales are moderately correlated with each other (r = .56, p < .001) and are strongly related to time spent in nature with large effect sizes (eta2 > .20).
Change in Exercise Goal Setting | pre and post 12-week intervention
  The SCT mechanism of goal setting will be measured using the Exercise Goal Setting Scale, a 10-item self-report 5pt Likert scale assessing goal-setting strategies such as self-monitoring and problem solving. Participants respond on a 5-point scale ranging from 1 (does not describe me) to 5 (completely describes me) and scores are averaged across the 10 items. This scale has good internal consistency (0.89).
Change in Support and Exercise | pre and post 12-week intervention
  Social support for exercise will be measured using a modified scale consisting of the Social Support and Exercise Survey, a 13-item survey that assess respondents' perceptions of positive and negative social support for exercise habits. Participants will rate the frequency with which CPSs and peers have done or said what was described in the items during the previous 3 months on a 5-point scale, ranging from 1 (none) to 5 (very often). Two subscales will be calculated (participation, rewards and punishments) for CPSs and peers with SMI. Cronbach's alphas range from .73-.80 in people with SMI. Research has shown that social support relates to goal setting practices in people with mental illness (r2=.11).
Physical Activity Participation | Ongoing during the 12-week intervention period
  Moderate to vigorous (MVPA) minutes per week will be objectively measured using Fitbit wearable devices (San Francisco, CA). Fitbit devices track a variety of health and fitness-related outcomes including steps, distance, heart rate, active minutes, calories, and sleep. Fitbit devices have high validity and reliability (ICCs range from 0.71-1.00 across studies)207-209 and have established feasibility and acceptability among adults with SMI. PA will be calculated as mean minutes of MVPA per session and per week. We will also assess physical activity using the Rapid Assessment of Physical Activity (RAPA). The RAPA is a 9-item dichotomous (Yes/No) measure of PA intensity (light, moderate, vigorous) and type (aerobic, flexibility, strength).
Change in Aerobic Fitness | pre and post 12-week intervention
  Aerobic fitness will be measured as distance traveled during a 6-minute walk test. Greater distance indicates better fitness.

OTHER OUTCOMES:
Feasibility - Facility | After completion of all waves of the study (approximately 2 years)
  Feasibility will be assessed via the Structured Assessment of FEeasibility (SAFE) which measures intervention feasibility within a mental health services framework. Completed by mental health facility administrators or staff, this measure includes 16 items that capture information in three categories: intervention, resource consequences, and evaluation. The SAFE measure has demonstrated excellent inter-rater and test-retest reliability (0.84, 95% confidence interval (CI) 0.79-0.89; 0.89, 95% CI 0.85-0.93 respectively). Rather than using a summary score, the individual items should be considered (e.g., yes, partial, no, unable to rate).
Change in Body Composition | pre and post 12-week intervention
  estimates include percent body fat via Tanita DC-430U or similar bioelectrical impedance scale, BMI via height and weight (via stadiometer and Tanita scale),waist circumference with spring-loaded Gulick tape measure
Change in Health-Related Quality of Life | pre and post 12-week intervention
  Health-related HRQOL will be assessed using the World Health Organization Quality of Life brief assessment (WHOQOL-BREF), a 26-item self-report questionnaire that measures four domains:
  physical health, psychological health, social relationships, and environment
Change in Depressive Symptoms | pre and post 12-week intervention
  Depressive symptoms will be assessed using an eight-item Personal Health Questionnaire depression scale (PHQ-9) a 9-item self-report scale which captures the severity of depressive symptoms experienced over the previous two weeks. We will also measure cross-cutting symptoms via DSM-5 (self-report, 23-items, 4pt Likert scale)
Change in Anxiety | pre and post 12-week intervention
  Measured via Generalized Anxiety Disorder (GAD-7; self-report, 7-items, 3pt Likert scale)
Change in General Health and Disability | pre and post 12-week intervention
  World Health Organization Disability Assessment Schedule (WHODAS 2.0; self-report, 12-items, 5pt Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Gina M Besenyi, MPH, PhD, Principal Investigator — Kansas State University
Locations (2):
- United States (2):
  - Serenity Behavioral Health Systems, Augusta, Georgia
  - Pawnee Mental Health, Junction City, Kansas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with colleagues who have a reasonable request and analysis plan with appropriate credit. Data will be shared according to NIMH's Data Sharing Policy (NOT-MH-19-033).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available to other interested researchers once major findings have been published or within two years of the project completion date, whichever is sooner.
Access Criteria: To be determined